CLINICAL TRIAL: NCT01406444
Title: IGF-1 and Bone Loss in Women With Anorexia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Karen Klahr Miller, MD, Chief, Neuroendocrine Unit, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2R01DK052625 (NIH)
Record Dates: First submitted 2011-07-26; First posted 2011-08-01 (Estimated); Results first posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Anorexia Nervosa; Osteopenia; Osteoporosis
Keywords: Anorexia Nervosa; Osteopenia; Osteoporosis; Bone density
MeSH Terms: conditions — Anorexia Nervosa; Bone Diseases, Metabolic; Osteoporosis | interventions — mecasermin; Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- rhIGF-1 followed by Risedronate (Active Comparator): Sequential therapy with rhIGF-1 (started at a dose of 30 mcg/kg subcutaneous BID and titrated) for 6 months followed by 6 months of risedronate 35mg PO once weekly
  Interventions: Drug: rhIGF-1; Drug: Risedronate
- Risedronate (Active Comparator): Risedronate 35mg PO once weekly for 12 months
  Interventions: Drug: Risedronate
- Placebo (Placebo Comparator): Placebo for 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: rhIGF-1 — Study participants will be started at a dose of 30 mcg/kg BID and will be titrated.
  Other Names: Increlex
  Arms: rhIGF-1 followed by Risedronate
Drug: Risedronate — Risedronate 35mg PO one time weekly
  Other Names: Actonel
  Arms: Risedronate; rhIGF-1 followed by Risedronate
Drug: Placebo — Placebo injections 30 mcg/kg BID, Placebo tablet PO once weekly
  Arms: Placebo

SUMMARY:
Anorexia nervosa is an eating disorder that can cause thinning of the bones (a decrease in bone density). A significant decrease in bone density is called osteopenia or osteoporosis. Sometimes the loss of bone density can be severe enough to cause breaks and fractures of the bones. It is not known what causes the bones to thin in anorexia nervosa. Women who have this condition often have thin or weak bones that are more likely to break. They also have very low levels of a chemical called IGF-1 in their body. This chemical is very important for increasing bone growth in puberty and for maintaining healthy adult bones. The investigators would like to find out if giving rhIGF-1 followed by risedronate or risedronate alone can lead to an increase in bone formation, bone density, and bone strength in women with anorexia nervosa.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years
* AN defined by DSM-IV diagnostic criteria, including weight less than 85% of ideal body weight (restricting or binge/purge type, BMI 15-17.5) OR meet criteria for sub-threshold AN, i.e., all DSM-IV criteria except that patients can have a BMI of <18.5 kg/m2 with or without amenorrhea
* Oral contraceptive use prior to enrollment
* BMD T score < -1.0
* Normal FSH and TSH or free T4
* Normal serum 25-OH vitamin D (>20 ng/mL) and calcium levels
* Ongoing care from a primary care provider
* Agree to use barrier contraception

Exclusion Criteria:

* Any subject with contraindications to risedronate
* Any subject with binge-purge subtype of anorexia nervosa who vomits regularly as their form of purging (vs. those who use laxatives or diuretics) and who have significant periodontal disease, tooth erosion or an invasive dental or periodontal procedure within the previous three months.
* Any disease known to affect bone, including untreated thyroid dysfunction, Cushing's or renal failure
* Any medication known to affect bone metabolism within 3 months of the study, excluding oral contraceptives. Bisphosphonates must have been discontinued for at least one year before participation
* Serum potassium <3.0 meq/L
* Serum ALT >3 times upper limit of normal
* eGFR of less than 30 ml/min
* Pregnant and/or breastfeeding
* Diabetes mellitus
* Active substance abuse, including alcohol
* History of malignancy
* Atraumatic fracture within the prior year

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2011-10; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Klibanski, MD, Principal Investigator — Massachusetts General Hospital; Erinne Meenaghan, NP, Study Chair — Massachusetts General Hospital; Karen Miller, MD, Study Director — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 148 subjects were consented and screened, 90 subjects were randomized, and 82 subjects completed the baseline visit. Of the 90 who were randomized, 8 subjects did not attend their scheduled baseline visits and did not receive study medication.
Period: Overall Study
Arm/Group | rhIGF-1 Followed by Risedronate | Risedronate | Placebo
Started | 33 | 33 | 16
Completed | 23 | 24 | 14
Not Completed | 10 | 9 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rhIGF-1 Followed by Risedronate | Risedronate | Placebo | Total
Number analyzed (Participants) | 33 | 33 | 16 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.9 (6.5) | 28.1 (7.1) | 25.4 (6.3) | 27.5 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 33 | 16 | 82
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 30 | 32 | 14 | 76
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 2 | 0 | 1 | 3
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 18.4 (1.5) | 18.4 (2.2) | 18.6 (1.7) | 18.4 (1.8)
Postero-anterior spine bone mineral density [Mean (Standard Deviation); unit: g/cm2] | 0.88 (0.12) | 0.86 (0.12) | 0.88 (0.12) | 0.88 (0.12)
Lateral spine bone mineral density [Mean (Standard Deviation); unit: g/cm2] | 0.67 (0.09) | 0.66 (0.09) | 0.67 (0.07) | 0.67 (0.09)

OUTCOME MEASURES:

1. Primary Outcome: Postero-anterior Spine Bone Mineral Density by DXA
Description: Postero-anterior spine bone mineral density by dual-energy X-ray absorptiometry
Time Frame: 12 Months
Measure: Least Squares Mean (Standard Error); unit: g/cm2
Arm/Group | rhIGF-1 Followed by Risedronate | Risedronate | Placebo
Number analyzed (Participants) | 23 | 24 | 14
g/cm2 | 0.891 (0.014) | 0.887 (0.014) | 0.874 (0.013)
Statistical Analysis 1: Comparison: rhIGF-1 Followed by Risedronate vs Placebo; Test type: Superiority; p = 0.03, Linear random effects model

2. Secondary Outcome: Lateral Spine Bone Mineral Density by DXA
Description: Lateral spine bone mineral density by dual-energy X-ray absorptiometry
Time Frame: 12 Months
Measure: Least Squares Mean (Standard Error); unit: g/cm2
Arm/Group | rhIGF-1 Followed by Risedronate | Risedronate | Placebo
Number analyzed (Participants) | 23 | 24 | 14
g/cm2 | 0.695 (0.012) | 0.677 (0.012) | 0.666 (0.010)
Statistical Analysis 1: Comparison: rhIGF-1 Followed by Risedronate vs Placebo; Test type: Superiority; p = 0.002, Linear random effects model
Statistical Analysis 2: Comparison: rhIGF-1 Followed by Risedronate vs Risedronate; Test type: Superiority; p = 0.04, Linear random effects model

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | rhIGF-1 Followed by Risedronate | Risedronate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33 | 0/16
Other Adverse Events (participants affected / at risk) | 19/33 | 18/33 | 5/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhIGF-1 Followed by Risedronate (N=33) | Risedronate (N=33) | Placebo (N=16)
Injection Site Irritation and/or Bruising (Skin and subcutaneous tissue disorders) | 15 (24) | 11 (14) | 2 (2) — Adverse event data collected at each study visit.
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (14) | 1 (1)
Upset Stomach (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Acid Reflux (Gastrointestinal disorders) | 4 (6) | 3 (4) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Headache (General disorders) | 1 (1) | 1 (1) | 2 (2)
Achiness (General disorders) | 1 (1) | 4 (5) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Dizziness (General disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-01-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT01406444/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT01406444/SAP_001.pdf